CLINICAL TRIAL: NCT02811523
Title: In Vivo Lung Perfusion (IVLP) as an Adjuvant Treatment for Patients Undergoing Surgical Resection of Pulmonary Metastases of Bone and Soft Tissues Sarcomas
Brief Title: In Vivo Lung Perfusion for Pulmonary Metastases of Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-8820
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Bone Sarcoma; Soft Tissue Sarcoma; Pulmonary Metastases
MeSH Terms: conditions — Bone Neoplasms; Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Doxorubicin 5 mcg/ml (Experimental): Doxorubicin 5mcg/ml by in vivo lung perfusion during surgical resection of pulmonary metastases
  Interventions: Drug: Doxorubicin
- Doxorubicin 7 mcg/ml (Experimental): Doxorubicin 7mcg/ml by in vivo lung perfusion during surgical resection of pulmonary metastases
  Interventions: Drug: Doxorubicin
- Doxorubicin 9 mcg/ml (Experimental): Doxorubicin 9mcg/ml by in vivo lung perfusion during surgical resection of pulmonary metastases
  Interventions: Drug: Doxorubicin
- Doxorubicin 7 mcg/ml - expansion (Experimental): Expansion group at ideal dose
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin by In Vivo Lung Perfusion

SUMMARY:
Sarcoma which has spread to the lungs is most often treated with surgery. Even with surgery, most patients will not be cured and will die from their disease, probably because of small cancer cells that are present in the lungs at the time of surgery, but cannot be seen or detected. It is for this reason that we are looking for a better treatment. Giving chemotherapy after surgery is generally not recommended because it has significant side effects and no benefit has been proven.

This study is investigating a new technique for delivering chemotherapy directly into the lungs at the time of surgery. Delivering chemotherapy directly to the lungs could potentially kill any microscopic cancer cells that are present in the lungs at the time of surgery, while sparing other major organs in the body from the side effects of chemotherapy. This technique is called In Vivo Lung Perfusion (IVLP). This is a Phase I, non-randomized, dose escalation study that will act as a pilot study for a larger prospective, multicenter, controlled clinical trial. Patients who have bilateral disease will have one lung undergo IVLP and the other lung will remain untreated with the IVLP (the other lung will be treated as current standard of care - either surgery or radiation) as a control lung. The patients will undergo a posterolateral thoracotomy. Lung metastases will be identified by visualization or palpation. After surgical isolation of the lung by proximal control of pulmonary artery and veins, IVLP will be initiated. After 3 hours of IVLP, the lung metastases will be removed in the usual fashion. Patients will be cared for post-surgery according to institutional standards. The patients will be followed for up to 2 years. The primary endpoint is safety. Secondary endpoints include additional safety endpoints and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Soft Tissue or Osteogenic Sarcoma
* Presence of bilateral pulmonary metastases
* 3 or more lung lesions in total
* Age less than 65 years
* ECOG 0-2
* Absence of extra-pulmonary disease
* Contralateral disease amenable to surgery or radiation
* All lung lesions in the lung to be treated with IVLP can be resected with wedge or segmental resections (non-IVLP treated lung will be treated with radiation or surgery 4-12 weeks prior to IVLP)

Exclusion Criteria:

* Patient has previously received more than 450 mg of doxorubicin
* Left Ventricular Ejection Fraction <50%
* History of significant pulmonary disease or pneumonitis
* Pregnant or lactating females
* Age 65 years or older, or less than 18 years
* Inability to understand the informed consent process
* Hypersenstivity to doxorubicin
* Current participation in another therapeutic clinical trial
* Previous lung metastatectomy

Ages: 0 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Safety of IVLP at selected dose levels by acute lung injury findings | Up to 2 years
Maximal tolerated dose by using a titration design | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cypel, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No